CLINICAL TRIAL: NCT02943746
Title: Utilizing Targeted Fortification to Evaluate the Effects of a High Versus Standard Protein Diet on Linear Growth and Body Composition in Infants < 1000 g Birth Weight.
Brief Title: Targeted Protein Fortification in Extremely Low Birth Weight Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Amy Hair, Assistant Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-38611
Record Dates: First submitted 2016-09-27; First posted 2016-10-25 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Premature Infants
Keywords: Standard Protein Diet; High Protein Diet; Growth; Body Composition; Extremely Low Birth Weight; Human Milk Derived Fortifier; Protein; Targeted Fortification; Human Milk Diet; Prematurity
MeSH Terms: conditions — Premature Birth | interventions — Diet, High-Protein

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Standard Protein Diet) (Active Comparator): Infants will receive a standard feeding regimen which consists of mother's own milk or donor human milk (DHM) with DHM derived fortifier.
  Once daily, a 24 hour batch of human milk is prepared for each infant (standard practice). A 2.5 mL sample will be analyzed for calories, protein, fat, and carbohydrates. Based on the amount of protein in the milk, fortification of feeds with donor human milk derived fortifier will be adjusted to reach an average of 3.5 to 3.8 g/kg/day of protein. Data will be recorded for milk analysis, nutrition, and infant growth.
  The diet will be continued until approximately 35 to 36 weeks postmenstrual age at which point a DXA scan will be performed.
  A serum blood urea nitrogen and creatinine as well as serum calcium, phosphorus, and alkaline phosphatase when the DXA is performed.
  Anthropometrics: weekly weight, length, and head circumference by trained research nurse.
  Interventions: Dietary Supplement: Standard Protein Diet
- Intervention Group (High Protein Diet) (Experimental): The intervention group will receive the same standard feeding regimen with the addition of extra milk fortification to give a high protein diet.
  Human milk will be prepared and analyzed in the same method as the control group. Based on the amount of protein in the milk, fortification of feeds with donor milk derived fortifier will be adjusted to reach an average of 4.2 to 4.5 g/kg/day.
  The diet will be continued until approximately 35 to 36 weeks PMA at which point a DXA scan will be performed.
  Infants will have 3 sets of labs. A serum blood urea nitrogen and creatinine as well as serum calcium, phosphorus, and alkaline phosphatase when the DXA is performed.
  Anthropometrics: weekly weight, length, and head circumference by trained research nurse.
  Interventions: Dietary Supplement: High Protein Diet

INTERVENTIONS:
Dietary Supplement: Standard Protein Diet — Based on the amount of protein in the milk, fortification of feeds with donor milk derived fortifier will be adjusted to reach an average of 3.5 to 3.8 g/kg/day.
  Arms: Control Group (Standard Protein Diet)
Dietary Supplement: High Protein Diet — Based on the amount of protein in the milk, fortification of feeds with donor milk derived fortifier will be adjusted to reach an average of 4.2 to 4.5 g/kg/day.
  Arms: Intervention Group (High Protein Diet)

SUMMARY:
While new innovations in the care of extremely premature infants have led to decreased morbidity and mortality, poor postnatal growth remains as a major challenge. Early growth in the postnatal period influences neurodevelopmental and growth outcomes.

This proposed study will challenge current nutritional regimens for infants < 1000 g birth weight (BW) by providing an exclusive human milk based diet with a higher amount of protein based on individual caloric and protein analysis of human milk utilizing targeted fortification. The investigators will evaluate the effects of a high versus standard protein enteral diet on growth and body composition in infants < 1000 g BW.

There are no published studies evaluating the effect of an exclusive human milk protein diet on body composition in premature infants. Research has shown that infants who receive this diet achieve growth at targeted standards but body composition has not been evaluated. As an all human milk diet is well tolerated and associated with improved outcomes in the highest risk neonates, it is imperative to evaluate the benefits of a high protein exclusive human milk diet and the possible positive changes in body composition, specifically lean mass, in these infants.

Results from this proposed study will immediately influence current nutritional practices and will provide landmark information regarding targeted fortification with provision of adequate protein providing the most optimal body composition in the most fragile and vulnerable infants.

DETAILED DESCRIPTION:
Primary Objective: To evaluate the effects of a high versus standard protein enteral diet utilizing targeted fortification on linear growth in infants < 1000 g birth weight (BW).

Hypothesis 1: Infants who receive a high protein diet will have increased length velocity at 36 weeks postmenstrual age when compared to infants who receive a standard protein diet.

Secondary Objective: To evaluate body composition by total body dual energy x-ray absorptiometry (DXA) at 36 weeks postmenstrual age in infants < 1000 g BW who received a high or standard protein enteral diet.

Hypothesis 2: Infants who received a high protein diet will have greater fat-free mass (lean mass) compared to infants who received a standard protein diet.

Protein and energy are key nutrients for growth. A low protein intake or protein to energy ratio may lead to poor linear growth and excess fat accumulation. Studies suggest that preterm infants require a high protein to energy ratio to obtain catch up growth without excessive fat accretion and that growth should focus on length gain and lean body mass.

Macronutrient analysis of donor human milk shows that mean protein values are 1.16 g/dL which is similar to term milk composition. Mother's milk and donor human milk protein content varies and is often lower than expected values. Infants may not be receiving the full amount of calories and protein needed to support growth.

The investigators plan to challenge current nutritional regimens for infants < 1000 g BW by providing an enteral diet with a higher amount of protein based on individual caloric and protein analysis of human milk also known as targeted fortification.

Study Design:

Using a prospective randomized study design, infants 500-1000 g BW receiving an exclusive human milk protein-based diet will be identified after admission to the NICU. For infants that meet inclusion criteria, the parent/guardian will be approached about the study. After informed written parental consent is obtained, infants will be randomized to receive either a high protein or standard protein diet. The standard protein diet (control group) providing 3.5-3.8 g/kg/day of protein represents our current practices. The high protein diet (intervention group) will provide 4.2-4.5 g/kg/day.

Control group (standard protein diet) versus the intervention group (high protein diet):

In the control group (standard protein diet), infants will receive a standard feeding regimen which consists of mother's own milk or donor human milk with donor human milk derived fortifier.

Once daily, a 24 hour batch of human milk will be prepared for each infant (standard practice in the milk bank). A 2.5 mL sample from the batch of human milk will be analyzed for calories (reported in kcal/oz) and protein, fat, and carbohydrate (reported in g/dL). Based on the amount of protein in the milk, fortification of feeds with donor human milk derived fortifier will be adjusted to reach an average of 3.5 to 3.8 g/kg/day of protein.

The intervention group (high protein diet) will receive the same standard feeding regimen with the addition of extra milk fortification to give a high protein diet. Based on the amount of protein in the milk, fortification of feeds with donor human milk derived fortifier, the number will be adjusted to reach an average of 4.2 to 4.5 g/kg/day.

Data will be recorded for milk analysis, nutrition, and infant growth.

The diets will be continued until approximately 35 to 36 weeks postmenstrual age (PMA) at which point a DXA scan will be performed.

Infants will have 3 sets of labs for study purposes. A serum Blood Urea Nitrogen (BUN) and creatinine will be performed 2-3 days and then 1 week after goal protein is achieved. At the time of the DXA scan, a serum calcium, phosphorus, and alkaline phosphatase will be performed.

Anthropometrics: weekly weight, length, and head circumference by trained research nurse.

Human Milk Samples: A 2.5 mL sample from the batch of human milk will be analyzed using a milk analyzer. This analyzer uses a secondary method for measurements. It is calibrated with bias samples from primary methods.

Tests: DXA scan will be used to evaluate body composition and provide measures of bone mineral, lean and fat mass.

Labs: BUN; creatinine, calcium, phosphorus, and alkaline phosphatase will be obtained at the time of DXA scan to measure bone mineral status.

Sample Size:

Based on admission data from our institution, approximately 120 infants < 1000 grams are admitted to our NICU each year. A projected 50% of eligible subjects to enroll in the study. Recruitment goal is 50 subjects in each group (n=100) with an additional 10 subjects per group to account for drop out providing a total sample size of 120 infants. This would provide 89% statistical power to detect a 15% difference (hypothesized in infants who receive high protein) in length velocity at the (two sided) 5% significance level.

Study Population:

Infants will be recruited from Level 3 NICU (Texas Children's Hospital) which admits inborn premature infants and from Level 4 NICU (Texas Children's Hospital) which admits infants born at another institution. Infants from Level 4 will be recruited if they were transferred to Texas Children's Hospital within the first 24 hours of life and have received an exclusive human milk diet.

Enrolled infants will be randomized to either the (control group or intervention group). Infants are usually within a range of birth weights, gestational ages and ethnicity. Male and females are usually close to 50%. The investigators are not recruiting specific ethnicities or genders as part of the inclusion criteria.

Study Duration:

Infants will be in this study from the time of consent to 35 - 36 weeks postmenstrual age.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight 500-1000 grams
* Reasonable expectation of survival for study duration (36 weeks postmenstrual age)
* Achieve any enteral feedings by 14 days of life
* Born at our institution or transferred from another institution within the first 24 hours of life and receive an exclusive human milk protein diet (mother's milk supplemented with donor human milk and donor human milk derived fortifier)

Exclusion Criteria:

* Birth weight > 1000 grams
* Less than a reasonable expectation for survival for the study duration, enrolled in another clinical study that affects nutritional management
* Failure to achieve enteral feeds by 14 days of life
* Major congenital anomalies or clinically significant congenital heart disease, presence of intestinal perforation or Stage 2 NEC prior to tolerating fortified feeds
* Early transfer to a non-study institution
* Unable to participate in the study for any reason based on decision of study investigator

Min Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Linear growth measured using an premature infant length board | Weekly until 35-36 postmenstrual age (PMA)
  Linear growth will be measured in centimeters (cm) per week. An average weekly linear growth will be calculated for each patient over the study period.These values will be compared to published standards for age.

SECONDARY OUTCOMES:
Body composition measured by dual energy x-ray absorptiometry | Performed at 35-36 weeks postmenstrual age
  Body composition parameters including fat mass, fat-free mass, bone mineral content will be measured in each patient and the results will be compared to standards for age.

CONTACTS AND LOCATIONS:
Overall Officials: Amy B Hair, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine / Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hair AB, Peluso AM, Hawthorne KM, Perez J, Smith DP, Khan JY, O'Donnell A, Powers RJ, Lee ML, Abrams SA. Beyond Necrotizing Enterocolitis Prevention: Improving Outcomes with an Exclusive Human Milk-Based Diet. Breastfeed Med. 2016 Mar;11(2):70-4. doi: 10.1089/bfm.2015.0134. Epub 2016 Jan 20. PMID 26789484
- [Background] Hair AB, Blanco CL, Moreira AG, Hawthorne KM, Lee ML, Rechtman DJ, Abrams SA. Randomized trial of human milk cream as a supplement to standard fortification of an exclusive human milk-based diet in infants 750-1250 g birth weight. J Pediatr. 2014 Nov;165(5):915-20. doi: 10.1016/j.jpeds.2014.07.005. Epub 2014 Aug 15. PMID 25130571
- [Background] Hair AB, Hawthorne KM, Chetta KE, Abrams SA. Human milk feeding supports adequate growth in infants </= 1250 grams birth weight. BMC Res Notes. 2013 Nov 13;6:459. doi: 10.1186/1756-0500-6-459. PMID 24220185